CLINICAL TRIAL: NCT06994286
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Pharmacokinetics, Safety, Tolerability and Pharmacodynamics of Single and Multiple Doses of MT-7117 in Chinese Healthy Subjects
Brief Title: The Purpose of This Study is to Investigate the Safety, Tolerability and Pharmacokinetics of MT-7117 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-7117-Z-104
Record Dates: First submitted 2025-04-24; First posted 2025-05-29 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Cohort A-1:MT-7117 100 mg (Active Comparator): single oral dose
  Interventions: Drug: MT-7117
- Cohort A-1:Placebo (Placebo Comparator): single oral dose
  Interventions: Drug: Placebo
- Cohort A-2:MT-7117 300mg (Active Comparator): single oral dose
  Interventions: Drug: MT-7117
- Cohort A-2:Placebo (Placebo Comparator): single oral dose
  Interventions: Drug: Placebo
- Cohort B-1:MT-7117 200mg (Active Comparator): single dose followed by once-daily oral dosing
  Interventions: Drug: MT-7117
- Cohort B-1:Placebo (Placebo Comparator): single dose followed by once-daily oral dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-7117 — Oral
  Other Names: Dersimelagon
  Arms: Cohort A-1:MT-7117 100 mg; Cohort A-2:MT-7117 300mg; Cohort B-1:MT-7117 200mg
Drug: Placebo — Oral
  Arms: Cohort A-1:Placebo; Cohort A-2:Placebo; Cohort B-1:Placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of MT-7117 in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male Chinese subjects or female Chinese subjects.
2. Subjects are aged 18 to 55 years, inclusive, at the time of informed consent.
3. Subjects must weigh at least 50 kg and have a body mass index (BMI) 19.0 to 26.0 kg/m2 both inclusive at Screening and Day -1.
4. Subjects must have acceptable clinical conditions in the opinion of the Investigator based upon the results of medical history, physical examination, clinical laboratory tests (biochemistry, hematology, coagulation, and urinalysis), vital signs and a 12-lead ECG at Screening and Day -1.
5. Subjects are able to provide written informed consent to participate in this study after reading Informed Consent Form (ICF), and after having the opportunity to discuss the study with the Investigator or designee.
6. In the Investigator's opinion, subjects are able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements.

Exclusion Criteria:

1. Subjects with presence and history of any clinically significant (in the opinion of the Investigator) cardiac, hepatobiliary, renal, gastrointestinal, respiratory, psychiatric/neurological, hematopoietic, endocrine, or skin disease.
2. Subjects with Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT) >=1.5 × upper limit of normal (ULN) and/or total bilirubin >ULN at Screening or Day -1.
3. Subjects who have a family history of long or short QT syndrome, hypokalemia, syncope, or Torsades de Pointes.
4. Subjects with clinically significant 12-lead ECG abnormalities or a QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 msec (male) and >470 msec (female), at Screening or Day -1.
5. Systolic blood pressure (SBP) outside the range of 90-140 mmHg, diastolic blood pressure (DBP) outside the range of 50-90 mmHg, or pulse rate outside the range of 50-100 bpm, taken in the sitting position at Screening or Day -1.
6. Presence or history of severe adverse reaction or allergy to any drug or food.
7. Donation or hemorrhage of 400 mL or more of blood within 12 weeks prior to Screening, or 200 mL or more of blood within 4 weeks prior to Screening.
8. Subjects who have a positive test for serologic reactions for syphilis, Hepatitis B surface (HBs) antigen, Hepatitis B core (HBc) antibody, Hepatitis C virus (HCV) antibody, or HIV antibody/antigen at Screening.
9. Presence or history of drug abuse, or a positive urine test for drugs of abuse at Screening or Day -1.
10. Presence or history (in the last two years) of alcohol abuse, or intake of more than 28 units/224 g of alcohol weekly for males or 21 units/168 g of alcohol weekly for females or a positive test for alcohol at Screening or Day -1. One unit/8 g is equivalent to a half-pint (280 mL) of beer or one measure (25 mL) of spirits or one glass (125 mL) of wine.
11. Subjects with presence or history of melanoma and/or presence or history of histologically confirmed dysplastic naevus.
12. Subjects with a first-degree relative with history of familial melanoma.
13. Subjects with Fitzpatrick skin type V or VI at Screening (only Part B).
14. Subjects who have suntanned using tanning beds, phototherapy, or artificial tanning products within 3 months prior to the Day -1. Sunburn due to sunlight may be included in the study if the Investigator judges that there is no problem with the study evaluation.
15. Subjects who used afamelanotide or melanotan within 6 months prior to the Day -1.
16. Subjects who used beta-carotene, or any other medications or supplements which may affect skin color, as judged by the Investigator within 3 months prior to Day -1.
17. Subjects who used any medication (including topical and herbal preparations) other than Investigational Medicinal Product (IMP) within 14 days (or 5 half-lives of the drug, whichever is longer) prior to the first dose of IMP.
18. Subjects who consumed any health food containing St John's Wort within 14 days prior to the first dose of IMP.
19. Subjects who consumed food or drink containing Seville oranges or grapefruit (including marmalade and fruit juices) within 7 days prior to the first dose of IMP.
20. Subjects who use tobacco or nicotine-containing products (snuff, chewing tobacco, cigarettes, cigars pipes, e-cigarettes, or nicotine replacement products) within 3 months prior to the first dose of IMP, or positive urine cotinine test at Screening or Day -1.
21. Subject who underwent surgery known to affect gastrointestinal absorption of the IMP (other than appendectomy and hernia repair/herniorrhaphy/hernioplasty).
22. Subjects who have participated in another clinical study involving blood sample collection or administration of IMP within 12 weeks prior to informed consent.
23. Subjects who have previously received MT-7117.
24. Female subjects who are pregnant (positive pregnancy test at Screening or Day -1) or lactating.
25. Male subjects and female subjects of childbearing potential who don't agree to use contraception as defined in the protocol.
26. Subjects the Investigator determined ineligible for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Time to maximum plasma concentration (tmax)of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Apparent plasma terminal elimination half-life (t1/2) of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Area under the plasma concentration-time curve from time zero to 24 hours (AUC0-24h) of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Area under the plasma concentration-time curve from time zero to 48 hours(AUC0-48h) of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-last) of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Area under the plasma concentration-time curve over the dosing interval (AUC0-τ) of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Area under the plasma concentration-time curve extrapolated from time zero to infinity (AUC0-∞). | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Terminal elimination rate constant (kel) of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Apparent oral clearance (CL/F) of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Apparent volume of distribution during the terminal phase after oral administration (Vz/F) of MT-7117 | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)
Mean residence time (MRT) of MT-7117. | PartA : pre-dose,0.5,3,4,5,6,8,12,24,48,96h post-dose, PartB : Day1,18(pre-dose,0.5,3,4,5,6,8,12h post-dose), Day2, Day3, Day5,6,8to12,14,16 (before IMP), Day19:24h*, Day20:48h*, Day21:72h* (*after last IMP)

SECONDARY OUTCOMES:
Number of subjects with Treatment-emergent Adverse events (AEs) (including serious AEs [SAEs] and hepatic AEs of special interest [AESIs]). | The time written informed consent is obtained from a subject until the end of the safety follow-up period or the withdrawal of the subject from the study (PartA), or until Day 21 or the withdrawal of the subject from the study (PartB).

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No